CLINICAL TRIAL: NCT05639686
Title: Comparison of Inhalational Anesthesia With Intravenous Tranexamic Acid and Total Intravenous Anesthesia on Surgical Field Quality in Endoscopic Sinus Surgery
Brief Title: TIVA vs TXA in Sinus Surgery to Evaluate Operative Blood Loss and Surgical Field Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Our Lady of the Lake Hospital (Other)
Collaborators: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Leslie Son, Research Scientist, Our Lady of the Lake Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TIVA vs TXA in Sinus Surgery
Record Dates: First submitted 2022-11-14; First posted 2022-12-06 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Rhinosinusitis Chronic; Sinus Cancer; Sinus Polyp; Encephalocele
MeSH Terms: conditions — Encephalocele | interventions — Tranexamic Acid; Propofol; Remifentanil

STUDY DESIGN:
Intervention Model Description: Double Blind, Randomized Cohort
Who Masked: Participant, Care Provider
Masking Description: The operating surgeon will be blinded to the type of anesthesia used by applying a surgical drape between surgeon and patient and anesthesia team. The patient will also not know which anesthesia arm they will be placed in as the randomization will occur prior to surgery and will only be known to the anesthesia team and other study team members who are not operating on the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Total Intravenous Anesthesia (TIVA) (Placebo Comparator): Patients will be induced with fentanyl 1-2µg/kg, propofol 2mg/kg, and lidocaine 1mg/kg. After orotracheal intubation, anesthesia will be maintained with propofol 150mg/kg/min, remifentanil 0.05-2µg/kg/min, and rocuronium or succinylcholine as indicated. This is standard of care for this procedure. Within 10 minutes of induction, patients in the control group will be administered a 100mL bolus of normal saline as placebo.
  Interventions: Drug: Total Intravenous Anesthesia
- Transexemic Acid (TXA) and Inhalational Anesthesia (Experimental): Patients will be induced with fentanyl 1-2µg/kg, propofol 2mg/kg, lidocaine 1mg/kg. After orotracheal intubation, anesthesia will be maintained with isoflurane 1.5-2% or sevoflurane 1-2%, as well as rocuronium or succinylcholine as indicated. Again standard of care procedure is applied. Within 10 minutes of induction, patients in the study group will be administered 15mg/kg TXA suspended in 100mL of normal saline intravenously.
  Interventions: Drug: Tranexamic acid injection; Drug: Inhalational isoflurane

INTERVENTIONS:
Drug: Tranexamic acid injection — Within 10 minutes of general anesthetic induction, 15mg/kg TXA suspended in 100mL of normal saline will be administered intravenously.
  Other Names: tranexamic acid (TXA)
  Arms: Transexemic Acid (TXA) and Inhalational Anesthesia
Drug: Total Intravenous Anesthesia — Within 10 minutes of induction, patients in the control (TIVA) group will be administered a 100mL bolus of normal saline as placebo.
  Other Names: total intravenous anesthesia (propofol, remifentanil)
  Arms: Total Intravenous Anesthesia (TIVA)
Drug: Inhalational isoflurane — Inhalational isoflurane or sevoflurane will be administered as a general anesthetic at the induction of the surgical procedure.
  Other Names: Inhalational anesthesia
  Arms: Transexemic Acid (TXA) and Inhalational Anesthesia

SUMMARY:
The goal of this interventional study is to compare the efficacy (surgical field quality and intra-operative blood loss) or cost of TIVA alone to general inhalational anesthetics with intravenous TXA in patient participants who are undergoing endoscopic sinus surgery.

The main questions the study aims to answer are:

* Is the surgical field quality better when using TIVA alone compared to general inhalational anesthetics with intravenous TXA?
* Is one method more financially advantageous to the participant and the institution compared to the other method?

Participants will be randomized into one of the two anesthesia cohorts prior to sinus surgery. One group will be given total intravenous anesthesia (TIVA) alone and the other will be given intravenous tranexamic acid (TXA) followed by general inhalational anesthesia.

Researchers will compare the TIVA group to the TXA group to see if one group exhibits a better surgery field viewing quality through a subjective evaluation and measurement of blood loss and also which anesthesia regimen is most cost effective upon conducting a cost analysis.

DETAILED DESCRIPTION:
This study aims to prospectively compare surgical field quality and intraoperative blood loss between patients treated with perioperative intravenous tranexamic acid (TXA) followed by general inhalational anesthesia (sevoflurane, isoflurane, or desflurane) to total intravenous anesthesia (TIVA) alone, which consists of propofol and remifentanil. A secondary objective would be to perform a cost analysis between these two groups to determine whether one method is financially more advantageous than the other.

This study will be a prospective double-blinded randomized control trial consisting of patients undergoing endoscopic sinus surgery to assess intraoperative blood loss, surgical field quality, and cost of the medications administered. The control group will receive total intravenous anesthesia without tranexamic acid during surgery. The study group will receive preoperative tranexamic acid with general inhaled anesthetics during surgery (detailed below). Randomization will be conducted via a pre-determined permuted block system (e.g. AABB, ABAB, BBAA, AABB, etc, where A is TIVA and B is general inhalational anesthetics with preoperative TXA). Subjects who consent to participate will be assigned to the A or B arm depending on whichever arm is listed next in the order.

Subjects will be informed about the study and consented during pre-operative clinic visits. The patient consent and HIPAA authorization forms will be presented at that time where the subject can read about the study followed by any verbal conversation or questions needed between the subject and the study team. This will be done in a private patient room setting. The subject will be notified that participation in the study is completely voluntary and that their medical care will not be affected regardless of their decision to participate. Of note, if patients decline to participate, they will undergo general anesthesia using TIVA without TXA, as this is the standard choice at our institution. Subjects will not receive payment or compensation for their participation.

ELIGIBILITY:
Inclusion Criteria:

* adults (age ≥18 years)
* will undergo endoscopic sinus surgery at Our Lady of the Lake Regional Medical Center
* includes patients who are undergoing endoscopic sinus surgery for myriad of indications, such as chronic rhinosinusitis, sinonasal tumors, and encephalocele repairs.
* includes patients who undergo both complete functional endoscopic sinus surgery, or FESS (i.e maxillary antrostomy, sphenoethmoidectomy, and frontal sinusotomy), as well as those who are undergoing limited functional endoscopic sinus surgeries (i.e. anything less than a complete FESS).

Exclusion Criteria:

* <18 years of age
* history of bleeding or coagulation disorder
* currently receiving anticoagulation therapy
* underlying condition with increased risk of thrombosis (e.g. antiphospholipid syndrome),
* history of thromboembolic disorder
* history of chronic kidney disease
* known allergy to tranexamic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Surgical Field Quality | Field quality measured Every 30 minutes over 4.5 hours of time using the Boezaart grading system.
  Surgical field quality during surgery
Intraoperative Blood loss | Measured once at the conclusion of surgery by measuring the total amount of fluid in the suction canisters minus the total amount of irrigation used
  Intraoperative blood loss at completion of surgery

SECONDARY OUTCOMES:
Cost Effectiveness between TIVA and TXA | Analysis Within 1 year of the procedure
  Comparison of cost of medications used for the TIVA arm to the arm with general anesthetics and TXA will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Hernandez, MD, Principal Investigator — LSU Health Sciences Center
Locations (1):
- Our Lady of the Lake Hospital, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No